CLINICAL TRIAL: NCT03512353
Title: An Open-label Phase 2 Study of Carfilzomib Plus Dexamethasone To Assess Tolerability and Adherence in Subjects With Relapsed or Refractory Multiple Myeloma at US Community Oncology Centers
Brief Title: A Study of Carfilzomib Plus Dexamethasone in Adults With Relapsed or Refractory Multiple Myeloma at US Community Oncology Centers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170596
Record Dates: First submitted 2018-04-02; First posted 2018-04-30 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Dexamethasone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib Plus Dexamethasone (Experimental): Participants received carfilzomib administered as an intravenous (IV) infusion twice-weekly for up to six 28-day cycles followed by once-weekly for another six 28-day cycles. The carfilzomib dose was 20 mg/m² on days 1 and 2 of cycle 1, 56 mg/m² for the remaining days of cycle 1 (days 8, 9, 15, and 16) and then on days 1, 2, 8, 9, 15, and 16 of each cycle for cycles 2 to 6, and 70 mg/m² on days 1, 8, and 15 of each cycle for cycles 7 to 12.
  Participants also received dexamethasone either orally or by IV infusion at a dose of 20 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 of cycles 1 to 6 and at a dose 40 mg once daily on days 1, 8, 15 of cycles 7 to 12.
  Interventions: Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be taken orally or by IV infusion at a dose of 20 mg once-daily on days 1, 2, 8, 9, 15, 16, 22, and 23 of cycles 1-6, and at a dose 40 mg once-daily on days 1, 8, 15 of cycles 7-12.
Drug: Carfilzomib — Carfilzomib will be administered at 20 mg/m² on days 1 and 2 of the first cycle. After that, carfilzomib will be administered at 56 mg/m² on days 8, 9, 15, and 16 of the first cycle, and then on days 1, 2, 8, 9, 15, and 16 on each 28-day cycle for the cycles 2 through 6. Starting with cycle 7 through cycle 12, carfilzomib will be administered at 70 mg/m² on days 1, 8, and 15 of each 28-day cycle. All
  Other Names: Kyprolis®

SUMMARY:
The primary objective was to describe the safety profile of carfilzomib plus dexamethasone regimen in adults with relapsed or refractory multiple myeloma (RRMM) with 1 to 3 prior lines of therapy at study entry.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label study in adults with RRMM in US community oncology centers. Adults with 1-3 prior lines of therapy at study entry are eligible to be screened for participation. Patients refractory to their last line of treatment are eligible to participate as long as their last line of treatment did not include a proteasome inhibitor (PI). The study will consist of a screening period of up to 28 days for bone marrow assessments and up to 21 days for all other assessments, up to 12 cycles of treatment, and a 30-day safety follow-up period following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Males or females greater than or equal to 18 years of age.
* Relapsed MM after last treatment or refractory while receiving non-proteasome inhibitor therapy.
* Measurable disease with at least 1 of the following assessed within 21 days prior to enrollment:

  * Immunoglobulin G (IgG) MM: serum monoclonal protein (M-protein) level ≥ 1.0 g/dL
  * IgA, IgD, IgE multiple myeloma: serum M protein level ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg per 24 hours
  * In subjects without measurable serum or urine M-protein, serum free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1.
* Subjects must have at least partial response (PR) to at least 1 line of prior therapy.
* Subjects must have received at least 1 but not more than 3 prior lines of therapy for MM (induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 line of therapy).
* Prior therapy with a proteasome inhibitor (PI) is allowed as long as the subject had at least a PR to most recent therapy with PI, was not removed due to toxicity (except for neuropathy), did not relapse within 60 days from discontinuation of PI, and will have at least a 6-month PI treatment-free interval from last dose received until enrollment. (Subjects may receive maintenance therapy with drugs that are not PI during this 6-month PI treatment-free interval).

Exclusion Criteria:

* Waldenström macroglobulinemia.
* Multiple myeloma of IgM subtype.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* History of plasma cell leukemia.
* Primary amyloidosis (patients with multiple myeloma with asymptomatic deposition of amyloid plaques found on biopsy would be eligible if all other criteria are met).
* Subjects with nephrotic range proteinuria (greater than or equal to 3 g albumin for 24 hours urine OR greater than or equal to 2 g albumin/1 g of creatinine on a random urine specimen).
* Myelodysplastic syndrome.
* History of other malignancy within the past 5 years, with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for greater than or equal to 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
  * Treated medullary or papillary thyroid cancer.
  * Similar neoplastic conditions with an expectation of greater than 95% five-year disease-free survival.
* Known human immunodeficiency virus (HIV) infection, hepatitis C infection (subjects with hepatitis C that achieve a sustained virologic response following antiviral therapy are allowed), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody that achieve sustained virologic response with antiviral therapy directed at hepatitis B are allowed).
* Acute or chronic graft-versus-host disease (any grade).
* Acute active infection requiring systemic antibiotics, antifungal, antiviral (except antiviral therapy directed at hepatitis B) agents within 14 days prior to enrollment.
* Known cirrhosis.
* Significant neuropathy (grades 3 to 4, or grade 2 with pain) within 14 days prior to enrollment.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment.
* Uncontrolled hypertension, defined as an average systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg. Subjects with controlled hypertension are eligible.
* Hepatic dysfunction within 21 days prior to enrollment: bilirubin 1.5 times the upper limit of normal (ULN) aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 3 times the ULN
* Active congestive heart failure with or without reduced ejection fraction (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT interval (QTc) of greater than 470 msec, pericardial disease, myocardial infarction within 4 months prior to enrollment.
* Known chronic obstructive pulmonary disease.
* Known interstitial pneumonitis.
* Immunotherapy within 21 days prior to enrollment.
* Chemotherapy with approved anticancer therapeutic within 21 days prior to enrollment.
* Glucocorticoid therapy (prednisone greater than 30 mg/day or equivalent) within 14 days prior to enrollment.
* Focal radiation therapy within 7 days prior to enrollment. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to enrollment (ie, prior radiation must have been to less than 30% of the bone marrow).
* Major surgery (except kyphoplasty) within 28 days prior to enrollment.
* Autologous or allogeneic stem cell transplant within 90 days prior to enrollment.
* Contraindication to dexamethasone.
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib).
* Intolerance to intravenous (IV) hydration.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Hepatic dysfunction within 21 days prior to enrollment: bilirubin greater than or equal to 1.5 times the upper limit of normal (ULN); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to 3 times the ULN.
* Left ventricular ejection fraction less than 40% assessed by transthoracic echocardiogram.
* Severe valvular disease assessed by transthoracic echocardiogram.
* Severe right-ventricular dysfunction assessed by transthoracic echocardiogram.
* Right-ventricular systolic pressure greater than 40 mm Hg assessed by transthoracic echocardiogram.
* Screening absolute neutrophil count (ANC) should be independent of growth factor support for greater than or equal to 1 week.
* Hemoglobin less than 80 g/L within 21 days prior to enrollment. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed, however most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin.
* Platelet count < 50 x 10^9/L (≤ 30 x 10^9/L if myeloma involvement in the bone marrow is > 50%) within 21 days prior to enrollment. Subjects should not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count.
* Estimated glomerular filtration rate (GFR) less than 30 mL/min/1.73 m^2 (per the Chronic Kidney Disease Epidemiology Collaboration formula) within 21 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (29):
- United States (29):
  - Research Site, Palm Springs, California
  - Research Site, Riverside, California
  - Research Site, Glenwood Springs, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Orange City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, River Forest, Illinois
  - Research Site, Tinley Park, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Paducah, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Midland, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Lincoln, Nebraska
  - Research Site, Florham Park, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Zanesville, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Corpus Christi, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Fredericksburg, Virginia
  - Research Site, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in the United States.
Period: Overall Study
Arm/Group | Carfilzomib Plus Dexamethasone
Started | 7
Received Treatment | 6
Completed (Study completion is defined as participants who received 12 cycles of treatment and completed the safety follow-up visit.) | 3
Not Completed | 4
Not completed — Sponsor Decision | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all enrolled participants who received at least 1 dose of any study treatment (ie, carfilzomib or dexamethasone).
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 4
  65 - 74 years | 1
  ≥ 75 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 5
Eastern Cooperative Oncology Group (ECOG) Performance Scale [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  Participants
    0 (Fully active) | 5
    1 (Restricted but ambulatory) | 1
    2 (Ambulatory but unable to work) | 0
Number of Prior Treatment Regimens [Count of Participants; unit: Participants]
  1 prior regimen | 4
  2 prior regimens | 1
  3 prior regimens | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed 12 Cycles of Treatment
Time Frame: 12 cycles (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Participants | 3

2. Primary Outcome: Percentage of Expected Dose of Carfilzomib Received in Cycles 1 to 12
Description: Percentage of expected dose of carfilzomib is defined as the percentage of actual cumulative dose (mg/m²) received by the participant relative to the full intended cumulative dose (mg/m²).
Time Frame: Up to 12 cycles (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Mean (Standard Deviation); unit: percentage of expected dose
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of expected dose | 90.53 (9.70)

3. Primary Outcome: Relative Dose Intensity of Carfilzomib in Cycles 1 to 12
Description: Relative dose intensity = actual dose intensity / planned dose intensity * 100, where dose intensity is the cumulative dose (mg) divided by the duration of the study drug administration (weeks).
Time Frame: Up to 12 Cycles (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Mean (Standard Deviation); unit: percentage of dose intensity
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of dose intensity | 89.85 (11.16)

4. Primary Outcome: Number of Participants With Carfilzomib Dose Modifications During Cycles 1 to 12
Description: Dose modification includes dosage adjustments, delays or discontinuations. A participant is counted only once for a reason category if there were multiple occurrences for the same reason. Participants may be counted in more than one category.
Time Frame: Cycles 1 - 12 (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Participants
  Any dose modification | 6
  Due to adverse event | 3
  Due to dose administration error | 1
  Per protocol | 1
  Due to weight change | 2
  Due to scheduling issues | 5

5. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events are defined as any adverse event with an onset date from the first dose through 30 days after the last dose of any study drug.
  Treatment-emergent related adverse events are adverse events considered related to at least one study drug by the investigator.
  Adverse events were graded using Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03, where Grade 1: Mild (asymptomatic or mild symptoms) Grade 2: Moderate (minimal, local or noninvasive intervention indicated) Grade 3: Severe (severe) or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated) Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: From the first dose of study drug until 30 days after the last dose (12 months)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Participants
  Any adverse event | 6
  Adverse events ≥ Grade 3 | 4
  Serious adverse events | 3
  Leading to discontinuation of carfilzomib | 0
  Leading to discontinuation of dexamethasone | 0
  Fatal adverse events | 1
  Treatment-related adverse events | 6
  Treatment-related adverse events ≥ Grade 3 | 4
  Treatment-related serious adverse events | 3
  Treatment-related fatal adverse events | 1

6. Secondary Outcome: Percentage of Expected Dose of Carfilzomib Received in Cycles 1 to 6 and 7 to 12
Description: as for outcome 2
Time Frame: Cycles 1-6 and 7-12 (each cycle is 28 days)
Population: All enrolled and treated participants with available data in each time period
Measure: Mean (Standard Deviation); unit: percentage of expected dose
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of expected dose
  Cycles 1 - 6 | 92.07 (8.70)
  Cycles 7 - 12: number analyzed (Participants) | 5
  Cycles 7 - 12 | 85.96 (12.98)

7. Secondary Outcome: Relative Dose Intensity of Carfilzomib in Cycles 1 to 6 and 7 to 12
Description: as for outcome 3
Time Frame: Cycles 1 - 6 and 7 - 12 (each cycle is 28 days)
Population: All enrolled and treated participants with available data in each time period
Measure: Mean (Standard Deviation); unit: percentage of dose intensity
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of dose intensity
  Cycles 1 - 6 | 92.80 (7.39)
  Cycles 7 - 12: number analyzed (Participants) | 5
  Cycles 7 - 12 | 85.96 (12.98)

8. Secondary Outcome: Number of Participants With Carfilzomib Dose Modifications During Cycles 1 to 6
Description: as for outcome 4
Time Frame: Cycles 1 - 6 (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Participants
  Any dose modification | 6
  Due to adverse event | 2
  Due to dose administration error | 1
  Per protocol | 1
  Due to weight change | 2
  Due to scheduling issues | 5

9. Secondary Outcome: Number of Participants With Carfilzomib Dose Modifications During Cycles 7 to 12
Description: as for outcome 4
Time Frame: Cycles 7 - 12 (each cycle is 28 days)
Population: Enrolled participants who received treatment during cycles 7 - 12
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 5
Participants
  Any dose modification | 4
  Due to adverse event | 3
  Due to scheduling issues | 1

10. Secondary Outcome: Number of Participants Who Discontinued Carfilzomib in Cycles 1 to 6 and 7 to 12
Description: Treatment discontinuation for all reasons in cycles 1 - 6 and cycles 7 - 12
Time Frame: Cycles 1 - 6 and 7 - 12 (each cycle is 28 days)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
Participants
  Discontinued during cycles 1 - 6 | 1
  Discontinued during cycles 7 - 12: number analyzed (Participants) | 5
  Discontinued during cycles 7 - 12 | 2

11. Secondary Outcome: Change From Baseline to Last Cycle of Treatment in European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire (EORTC QLQ)-Core 30 (C30)
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) is a 30-item questionnaire used to assess the overall quality of life in cancer patients. EORTC QLQ-C30 was administered on day 1 of each treatment cycle. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  For each of these scales, scores range from 0 to 100. For the GHS and 5 functional scales a high score indicates better global health status/functioning and a positive change from baseline indicates improvement. For the 9 symptom scales, a high score indicates a higher level of symptoms, and a negative change from Baseline indicates an improvement in symptoms.
Time Frame: Baseline (cycle 1 day 1) to cycle 12 day 1
Population: All enrolled and treated participants
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
scores on a scale
  Physical Functioning | -15.6 (15.6)
  Role Functioning | -16.7 (25.8)
  Emotional Functioning | -5.6 (15.5)
  Cognitive Functioning | 2.8 (12.6)
  Social Functioning | -19.4 (19.5)
  Fatigue | 9.3 (10.9)
  Pain | -8.3 (25.3)
  Nausea and Vomiting | 0.0 (10.5)
  Global Health Status | -5.6 (10.1)
  Dyspnoea | 22.2 (27.2)
  Appetite Loss | 5.6 (13.6)
  Insomnia | -5.6 (13.6)
  Constipation | 11.1 (27.2)
  Diarrhoea | -5.6 (25.1)
  Financial Difficulties | 5.6 (13.6)

12. Secondary Outcome: Change From Baseline in Average EORTC QLQ-C30 Scores During Cycles 2 to 6 in Participants Who Completed 12 Cycles of Treatment
Description: EORTC QLQ-C30 was administered on day 1 of each treatment cycle. EORTC QLQ-C30 is a 30-item questionnaire used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  For each of these scales, scores range from 0 to 100. For the GHS and 5 functional scales a high score indicates better global health status/functioning and a positive change from baseline indicates improvement. For the 9 symptom scales, a high score indicates a higher level of symptoms, and a negative change from Baseline indicates an improvement in symptoms.
  Change from baseline is the difference in the average score from cycles 2 to 6 and the score on cycle 1 day 1.
Time Frame: Baseline (cycle 1 day 1) and cycles 2 - 6
Population: Enrolled participants who completed 12 cycles of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 3
scores on a scale
  Physical Functioning | -16.9 (10.2)
  Role Functioning | -7.8 (18.4)
  Emotional Functioning | -13.9 (19.5)
  Cognitive Functioning | -4.4 (23.7)
  Social Functioning | -12.2 (15.8)
  Fatigue | 11.9 (9.0)
  Pain | -3.3 (20.8)
  Nausea and Vomiting | 10.0 (5.8)
  Global Health Status | -9.4 (9.5)
  Dyspnoea | 8.9 (7.7)
  Appetite Loss | 13.3 (13.3)
  Insomnia | -11.1 (3.9)
  Constipation | -4.4 (20.4)
  Diarrhoea | -2.2 (16.8)
  Financial Difficulties | 6.7 (24.0)

13. Secondary Outcome: Change From Cycle 7 Day 1 in Average EORTC QLQ-C30 Scores During Cycles 8 to 12 in Participants Who Completed 12 Cycles of Treatment
Description: EORTC QLQ-C30 was administered on day 1 of each treatment cycle. EORTC QLQ-C30 is a 30-item questionnaire used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  For each of these scales, scores range from 0 to 100. For the GHS and 5 functional scales a high score indicates better global health status/functioning and a positive change from baseline indicates improvement. For the 9 symptom scales, a high score indicates a higher level of symptoms, and a negative change from baseline indicates an improvement in symptoms.
  Change was calculated as the difference in the average score from cycles 8 to 12 and the score on cycle 7 day 1.
Time Frame: Cycle 7 day 1 and cycles 8 - 12
Population: Enrolled participants who completed 12 cycles of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 3
scores on a scale
  Physical Functioning | 6.2 (5.6)
  Role Functioning | -1.1 (5.1)
  Emotional Functioning | 1.1 (1.9)
  Cognitive Functioning | 13.3 (12.0)
  Social Functioning | 0.0 (6.7)
  Fatigue | 6.7 (16.0)
  Pain | 13.3 (12.0)
  Nausea and Vomiting | 6.7 (8.8)
  Global Health Status | 2.2 (1.9)
  Dyspnoea | 22.2 (13.9)
  Appetite Loss | 4.4 (7.7)
  Insomnia | 4.4 (7.7)
  Constipation | 0.0 (20.0)
  Diarrhoea | -2.2 (10.2)
  Financial Difficulties | -4.4 (3.9)

14. Secondary Outcome: Change From Baseline to Last Cycle of Treatment in EORTC QLQ Multiple Myeloma Module (MY-20) Scores
Description: EORTC QLQ-MY20 is a 20-item questionnaire used in clinical research to assess health-related quality of life in multiple myeloma patients. Questions are answered on a 4-point scale from 1 'Not at All' to 4 'Very Much'.
  The QLQ-MY20 includes four domains (Disease Symptoms, Side-Effects of Treatment, Body Image and Future Perspective).
  Domain scores are calculated as averages and transformed to range from 0 to 100.
  For the Disease symptoms and side-effects of treatments scales a higher score represents a higher level of symptoms/problems and a negative change from baseline value indicates reduction (i.e. improvement) in symptoms. For the body image and future perspectives scales a higher score represents a higher level of functioning, and a positive change from baseline indicates improvement.
Time Frame: Baseline (cycle 1 day 1) and cycle 12 day 1
Population: All enrolled and treated participants
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
scores on a scale
  Disease Symptoms | -5.6 (17.9)
  Side-effects of Treatment | 6.5 (7.9)
  Body Image | -5.6 (13.6)
  Future Perspective | 1.9 (21.6)

15. Secondary Outcome: Change From Baseline in Average EORTC QLQ-MY20 Scores During Cycles 2 to 6 in Participants Who Completed 12 Cycles of Treatment
Description: EORTC QLQ-MY20 is a 20-item questionnaire used in clinical research to assess health-related quality of life in multiple myeloma patients. Questions are answered on a 4-point scale from 1 'Not at All' to 4 'Very Much'.
  The QLQ-MY20 includes four domains (Disease Symptoms, Side-effects of Treatment, Body Image and Future Perspective).
  Domain scores are calculated as averages and transformed to range from 0 to 100.
  For the disease symptoms and side-effects of treatment scales a higher score represents a higher level of symptoms/problems and a negative change from baseline value indicates reduction (i.e. improvement) in symptoms. For the body image and future perspectives scales a higher score represents a higher level of functioning, and a positive change from baseline indicates improvement.
  Change from baseline is the difference in the average score from cycles 2 to 6 and the score on cycle 1 day 1.
Time Frame: Baseline (cycle 1 day 1) and cycles 2 - 6
Population: Enrolled participants who completed 12 cycles of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 3
scores on a scale
  Disease Symptoms | -13.2 (16.4)
  Side-effects of Treatment | 10.6 (6.8)
  Body Image | -2.8 (4.8)
  Future Perspective | 6.1 (25.3)

16. Secondary Outcome: Change From Cycle 7 Day 1 in Average EORTC QLQ-MY20 Scores Over Cycles 8 to 12 in Participants Who Completed 12 Cycles of Treatment
Description: EORTC QLQ-MY20 is a 20-item questionnaire used in clinical research to assess health-related quality of life in multiple myeloma patients. Questions are answered on a 4-point scale from 1 'Not at All' to 4 'Very Much'.
  The QLQ-MY20 includes four domains (Disease Symptoms, Side- Effects of Treatment, Body Image and Future Perspective).
  Domain scores are calculated as averages and transformed to range from 0 to 100.
  For the disease symptoms and side effects of treatments scales a higher score represents a higher level of symptoms/problems and a negative change from baseline value indicates reduction (i.e. improvement) in symptoms. For the body image and future perspectives scales a higher score represents a higher level of functioning, and a positive change from baseline indicates improvement.
  Change was calculated as the difference in the average score from cycles 8 to 12 and the score on cycle 7 day 1.
Time Frame: Cycle 7 day 1 and cycles 8 - 12
Population: Enrolled participants who completed 12 cycles of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 3
scores on a scale
  Disease Symptoms | 8.2 (7.6)
  Side-effects of Treatment | -3.8 (3.8)
  Body Image | -17.8 (20.4)
  Future Perspective | 3.0 (7.1)

17. Secondary Outcome: Overall Response Rate (ORR)
Description: Disease response and progression were determined using International Myeloma Working Group Uniform Response Criteria (IMWG-URC) 2016, assessed by the Investigator. Per IMWG, determination of disease response requires: serum free light chain (SFLC), serum and urine protein electrophoresis (SPEP, UPEP, respectively), serum and urine immunofixation (SIFE, UIFE, respectively), bone marrow aspirate (for complete response confirmation), corrected calcium (cCa), and plasmacytoma evaluation, if present at screening.
  Best overall response is defined as a participant's best response during the study. Overall response rate is defined as the percentage of participants achieving a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: Disease assessments were performed every 28 days up to 12 months from enrollment.
Population: All enrolled and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of participants | 83.3 [35.9 to 99.6]

18. Secondary Outcome: Overall Response Rate (ORR) After 6 Cycles
Description: Disease response and progression were determined using International Myeloma Working Group Uniform Response Criteria (IMWG-URC) 2016, assessed by the Investigator. Per IMWG, determination of disease response requires: serum free light chain (SFLC), serum and urine protein electrophoresis (SPEP, UPEP, respectively), serum and urine immunofixation (SIFE, UIFE, respectively), bone marrow aspirate (for CR confirmation), corrected calcium, and plasmacytoma evaluation, if present at screening.
  Overall response rate after 6 cycles is defined as the percentage of participants achieving a best overall response during the first 6 treatment cycles of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: Disease assessments were performed every 28 days up to 6 cycles of treatment (each cycle was 28 days)
Population: All enrolled and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of participants | 83.3 [35.9 to 99.6]

19. Secondary Outcome: Overall Response Rate (ORR) by Prior Lines of Therapy
Description: Disease response and progression were determined using International Myeloma Working Group Uniform Response Criteria (IMWG-URC) 2016, assessed by the Investigator. Per IMWG, determination of disease response requires: serum free light chain (SFLC), serum and urine protein electrophoresis (SPEP, UPEP, respectively), serum and urine immunofixation (SIFE, UIFE, respectively), bone marrow aspirate (for CR confirmation), corrected calcium, and plasmacytoma evaluation, if present at screening.
  Best overall response is defined as a participant's best response during the study. Overall response rate is defined as the percentage of participants achieving a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: Disease assessments were performed every 28 days up to 12 months from enrollment.
Population: All enrolled and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 1 Prior Line of Therapy: Participants with 1 prior line of therapy for multiple myeloma.
- 2+ Prior Lines of Therapy: Participants with ≥ 2 prior lines of therapy for multiple myeloma.
Arm/Group | 1 Prior Line of Therapy | 2+ Prior Lines of Therapy
Number analyzed (Participants) | 4 | 2
percentage of participants | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0]

20. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) Events at 12 Months
Description: Progression-free survival events include disease progression or death due to any cause.
  Disease progression was determined by the Investigator according to IMWG criteria.
Time Frame: 12 months
Population: All enrolled and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib Plus Dexamethasone
Number analyzed (Participants) | 6
percentage of participants | 50.0

21. Secondary Outcome: Percentage of Participants With PFS Events by Prior Lines of Therapy
Description: Progression-free survival (PFS) events include disease progression or death due to any cause.
  Disease progression was determined by the Investigator according to IMWG criteria.
Time Frame: Disease assessments were performed every 28 days up to 12 months from enrollment.
Population: All enrolled and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | 1 Prior Line of Therapy | 2+ Prior Lines of Therapy
Number analyzed (Participants) | 4 | 2
percentage of participants | 50.0 | 50.0

ADVERSE EVENTS:
Time Frame: All cause mortality - from enrollment to end of study (13 months) Adverse Events - From the first dose of study drug until 30 days after the last dose (12 months)
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Carfilzomib Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib Plus Dexamethasone (N=6)
Cardiac arrest (Cardiac disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib Plus Dexamethasone (N=6)
Anaemia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dizziness exertional (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Because of the limited sample size, no meaningful conclusions on the study objectives can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03512353/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03512353/SAP_001.pdf